CLINICAL TRIAL: NCT03558620
Title: Effect of an Endoscopic Bite Block on Mask Ventilation in Anesthetized and Paralyzed Patients
Brief Title: Effect of an Endoscopic Bite Block on Mask Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jin-Young Hwang, Associate professor, Department of Anesthesiology and Pain medicine, SMG-SNU Boramae Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2018/00/0000
Record Dates: First submitted 2018-04-26; First posted 2018-06-15 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Ventilator Lung
Keywords: manual ventilation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group 1O2 (Experimental): A fitting mask is held by one hand -> one hand with an endoscopic bite block -> held by two hands
  Interventions: Procedure: mask ventilation
- Group 12O (Experimental): A fitting mask is held by one hand -> held by two hands-> one hand with an endoscopic bite block
  Interventions: Procedure: mask ventilation
- Group O12 (Experimental): A fitting mask is held by one hand with an endoscopic bite block->by one hand -> by two hands
  Interventions: Procedure: mask ventilation
- Group O21 (Experimental): A fitting mask is held by one hand with an endoscopic bite block -> by two hands-> one hand
  Interventions: Procedure: mask ventilation
- Group 21O (Experimental): A fitting mask is held by two hands -> one hand -> one hand with an endoscopic bite block
  Interventions: Procedure: mask ventilation
- Group 2O1 (Experimental): A fitting mask is held by two hands ->one hand with an endoscopic bite block-> by one hand
  Interventions: Procedure: mask ventilation

INTERVENTIONS:
Procedure: mask ventilation — mask ventilation (one-handed ventilation, one-handed with an endoscopic bite block, and two-handed ventilation)

SUMMARY:
Evaluation of effects of an endoscopic bite block on mask ventilation. In the present study, expiratory tidal volume and minute ventilation are measured under same pressure controlled mode in ventilator with three kinds of holding a mask. ( by one hand, one hand with an endoscopic bite block and two hand hold.)

DETAILED DESCRIPTION:
Evaluation of effects of an endoscopic bite block on mask ventilation. In the present study, expiratory tidal volume and minute ventilation are measured under the same pressure controlled mode in ventilator (Pressure 15cmH2O, Respiratory rate 15/min, I:E=1:1) with three kinds of holding a mask. ( by one hand, one hand with an endoscopic bite block and two hand hold.)

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for elective surgery under general anesthesia and agree with the purpose of the study

Exclusion Criteria:

* patients with diseases or structural abnormalities in the upper airway, wobbly teeth, and limited mouth opening of less than 3.5 cm or those who were at risk of aspiration

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2018-12-12 (Actual)

PRIMARY OUTCOMES:
Expiratory tidal volume | during mask ventilation after anesthesia induction
  Expiratory tidal volume with one-hand mask ventilation, one-handed mask ventilation with an endoscopic bite block, and two-handed ventilation

SECONDARY OUTCOMES:
Minute ventilation | during mask ventilation after anesthesia induction
  Minute ventilationwith one-hand mask ventilation, one-handed mask ventilation with an endoscopic bite block, and two-handed ventilation
Incidence of inadequate ventilation or dead space ventilation | during mask ventilation after anesthesia induction
  Inadequate mask ventilation and dead-space ventilation are defined as a mean expiratory tidal volume of less than 4 mL kg-1 of predicted body weight and a mean expiratory tidal volume of less than 150 mL per breath with no clinical signs, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Young Hwang, M.D., phD, Principal Investigator — Seoul Metropolitan Government Seoup National University Boramae Medical Center
Locations (1):
- Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hart D, Reardon R, Ward C, Miner J. Face mask ventilation: a comparison of three techniques. J Emerg Med. 2013 May;44(5):1028-33. doi: 10.1016/j.jemermed.2012.11.005. Epub 2013 Mar 7. PMID 23473817
- [Background] Joffe AM, Hetzel S, Liew EC. A two-handed jaw-thrust technique is superior to the one-handed "EC-clamp" technique for mask ventilation in the apneic unconscious person. Anesthesiology. 2010 Oct;113(4):873-9. doi: 10.1097/ALN.0b013e3181ec6414. PMID 20808210
- [Background] Walsh JH, Maddison KJ, Platt PR, Hillman DR, Eastwood PR. Influence of head extension, flexion, and rotation on collapsibility of the passive upper airway. Sleep. 2008 Oct;31(10):1440-7. PMID 18853942